CLINICAL TRIAL: NCT04715555
Title: SAFER Wearables Study: A Study of the Acceptability and Performance of Wearables for Atrial Fibrillation Screening in Older Adults
Brief Title: A Study of the Acceptability and Performance of Wearables for Atrial Fibrillation Screening in Older Adults
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: City, University of London (Other); University of Leicester (Other)
Responsible Party: Principal Investigator, Peter Charlton, British Heart Foundation Research Fellow, University of Cambridge
Other Study IDs: IRAS 283812; FS/20/20/34626 (Other Grant/Funding Number: British Heart Foundation); 20/EM/0255 (Other: REC reference)
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation; Paroxysmal Atrial Fibrillation
Keywords: Wearable Electronic Devices; Electrocardiography, Ambulatory; Photoplethysmography; Arrhythmias, Cardiac; Diagnostic Screening Programs; Ergonomics
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Atrial Fibrillation: Participants with a diagnosis of atrial fibrillation (AF) who exhibited AF in previous AF screening (as part of the SAFER Programme).
  Interventions: Device: Electrocardiogram monitoring; Device: Electrocardiogram recording; Device: Photoplethysmogram monitoring; Other: Feedback questionnaire
- Non-Atrial Fibrillation: Participants without a diagnosis of atrial fibrillation (AF) who have previously undergone AF screening (as part of the SAFER Programme).
  Interventions: Device: Electrocardiogram monitoring; Device: Electrocardiogram recording; Device: Photoplethysmogram monitoring; Other: Feedback questionnaire

INTERVENTIONS:
Device: Electrocardiogram monitoring — Continuous monitoring using a wearable, single-lead electrocardiography (ECG) device affixed to the chest.
Device: Electrocardiogram recording — Intermittent electrocardiogram (ECG) recordings taken using a wearable device on the wrist.
Device: Photoplethysmogram monitoring — Photoplethysmogram monitoring using a wearable device on the wrist.
Other: Feedback questionnaire — A questionnaire to collect feedback on participants' experiences of wearing the devices.

SUMMARY:
--- Background and study aim

Atrial fibrillation (AF) is an irregular heart rhythm which causes a five-fold increase in the risk of stroke. Approximately one in ten people aged over 70 have AF. If AF is recognised then the risk of stroke can be reduced by taking tablets regularly. AF can be difficult to recognise as it can occur without symptoms and only intermittently. Consequently, AF is not recognised in many people, meaning they live with an increased risk of stroke. Therefore, it is important to find ways to identify AF more reliably.

Recently, wearable devices have been developed which could be useful for identifying AF. Several devices can monitor heart activity in daily life, including wristbands, smart watches and chest patch monitors. The aim of this study is to assess the acceptability and performance of wearables for use in AF screening in older adults.

The primary objective is to determine the feasibility of measuring inter-beat-intervals using a wristband. The secondary objectives are:

(i) to determine the acceptability of wearables; (ii) to determine the acceptability of the screening approach; (iii) to assess the performance of wearables for acquiring signals; (iv) to assess the performance of signal processing algorithms; and (v) to assess the performance of wearables for AF screening.

--- Who can participate?

Selected people who have previously participated in the SAFER Programme can participate in this study. The Investigators will invite previous SAFER Programme participants to also participate in this study, aiming to enrol 65 without AF, and 65 with AF.

--- What does the study involve?

Participants will be asked to wear three devices for seven days: Two wristbands (like watches), and one chest patch (like a plaster). These devices will collect measurements of their heart's activity. The Investigators will also ask participants to tell them how they found wearing the devices by completing a questionnaire. The Investigators will compare how participants found wearing each device, and how accurately each device identifies AF.

--- What are the possible benefits and risks of participating?

There will be no direct benefit to participants, although this research is intended to benefit future patients like them. Some participants may experience irritation or redness whilst wearing a chest patch - participants will be advised that if this occurs then they should remove it straightaway.

DETAILED DESCRIPTION:
--- Where is the study run from?

The University of Cambridge.

--- Study procedures

Participants will be asked to:

1. Consent: Participants will be asked to confirm their consent to take part by posting the enclosed consent form to the Investigators in a prepaid envelope.
2. Device delivery: The Investigators will send participants the devices, a detailed instruction leaflet, and a questionnaire.
3. Training: The Investigators will explain to participants how to wear and use the devices over the telephone, referring to the instruction leaflet.
4. Wear the devices: Participants will be asked to wear the devices for seven days, going about their daily life as normal. The devices are waterproof. If a participant has chest hair then they will need to shave a small area for the chest-patch to stick to. The Investigators will ask participants to use the watch four times each day to record heart activity for 30 seconds. Participants will be asked to plug in a small hub which will send information from the devices. The Investigators will telephone participants during the study to check for any problems.
5. Questionnaire: Participants will be asked to complete a questionnaire on the devices after wearing them.
6. Return devices: At the end, the Investigators will telephone participants and arrange a courier to pick up the devices and questionnaire from their home (which the Investigators will arrange and pay for).

Participants will be given an instruction leaflet with further details of each step.

ELIGIBILITY:
Inclusion Criteria:

* AF screening successfully completed during the SAFER Programme
* Aged 65 years or over
* Lives in private accommodation
* Willing and able to give informed consent

Exclusion Criteria:

* Regularly sleeps on front
* Has a chest wound
* Previous reaction to, or known allergy to ECG electrodes or silicone
* Receiving palliative care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Potential participants for the study will be identified from amongst previous participants of the SAFER Programme (ISRCTN 16939438 and ISRCTN 72104369).
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-05-23 (Estimated); Study Completion 2025-05-23 (Estimated)

PRIMARY OUTCOMES:
The performance of each wrist-worn wearable approach for identifying AF participants | 7 days
  Sensitivity and specificity

SECONDARY OUTCOMES:
The time for which participants report wearing the wearables | 7 days
  Duration of time, expressed as median (lower, upper quartiles)
The number of wrist-ECG recordings taken by participants | 7 days
  Median (lower, upper quartiles)
The proportion of participants in whom AF was observed, who recorded a wrist-ECG signal during an AF episode | 7 days
  Percentage
Participant-reported experiences of wearing the wearables | Day 8
  Feedback obtained from questionnaires (including some responses provided on a Likert Scale with options 'Strongly agree', 'Agree', 'Neither agree nor disagree', 'Disagree', and 'Strongly disagree').
Device packs lost in transit | Day 1, end of participation
  The number for both outward and return legs
The time for which each device attempts to record signals | 7 days
  The time from the wearable being first applied to the time of either it being finally removed, or its battery running out (whichever occurs first). Expressed as median (lower, upper quartiles)
The time for which wearable signals are acquired | 7 days
  Duration of time, and proportion of recording time, expressed as median (lower, upper quartiles). 'Wearable signal' is defined as a non-flat-line signal.
The proportion of recording time for which wearable signals are of high quality | 7 days
  Percentage, expressed as median (lower, upper quartiles)
The proportion of recording time for which high quality wearable signals are acquired at different times of day | 7 days
  Percentages, expressed as median (lower, upper quartiles)
The agreement between interbeat-intervals (IBIs) provided by IBI wristbands, and derived from reference ECG chest-patch signals | 7 days
  Limits of Agreement technique (consisting of the bias and limits of agreement)
The agreement between ECG features derived from wrist-ECGs and reference ECG chest-patch signals. | 7 days
  Limits of Agreement technique (consisting of the bias and limits of agreement)
The performance of an algorithm to detect AF from wrist-ECG signals | 7 days
  sensitivity and specificity
The performance of an algorithm to detect possible AF from IBI wristband signals | 7 days
  Sensitivity and specificity
The proportion of possible AF episodes detected from IBI wristband signals for which the reference ECG exhibited a verified AF episode lasting for ≥ 90 seconds from the start time of the possible episode | 7 days
  Percentage, expressed as median (lower, upper quartiles)
The agreement between AF burden estimates obtained from wrist devices and the reference ECG chest-patch | 7 days
  Limits of Agreement technique (consisting of the bias and limits of agreement)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Charlton, MEng, PhD, Principal Investigator — University of Cambridge
Locations (1):
- University of Cambridge, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The following data from individual participants will be anonymised and shared:
  * Participant characteristics
  * Quantitative questionnaire data (providing feedback on the wearable devices)
  * Device data including physiological signals, physiological parameters, and technical parameters.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be made available within 12 months of the study ending. It will made available indefinitely via an online repository.
Access Criteria: None planned